CLINICAL TRIAL: NCT04045158
Title: Diaphragm Ultrasound in Neuromuscular Disorders
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Principal Investigator, Abdallah FAYSSOIL, MD PhD, Centre d'Investigation Clinique et Technologique 805
Other Study IDs: DIAPH-NMD
Record Dates: First submitted 2019-07-22; First posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Muscular Dystrophies
Keywords: diaphragm; ultrasound; echocardiography
MeSH Terms: conditions — Muscular Dystrophies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Muscular dystrophies are neurologic disease with higher morbidity and mortality. Cardiac function and respiratory muscles can be affected, in addition with skeletal muscle deficiency . Lung function is classically assessed with functionnal pulmonary tests (FPT) . Ultrasound recently emerged as a non-invasive tool to assess diaphragm function.

The aims of the study are:

* to provide the spectrum of diaphragm ultrasound in patients with muscular dystrophies
* to assess the correlation between diaphragm ultrasound and FPT
* to assess the correlation between diaphragm ultrasound and cardiac function

ELIGIBILITY:
Inclusion Criteria:

* Duchenne muscular dystrophy,
* Becker muscular dystrophy,
* LGMD,
* myotonic dystrophy type 1 and type 2,
* metabolic myopathy,
* mitochondrial myopathy,
* FSHD1 and 2,
* myasthenia

Exclusion Criteria:

* history of cardiac surgery
* history of thoracic surgery
* brain traumatism

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with neuromuscular diseases admitted for a cardio-respiratory function evaluation
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-12-28 (Estimated); Study Completion 2020-05-10 (Estimated)

PRIMARY OUTCOMES:
diaphragm ultrasound motion | 1 year
  using echography

SECONDARY OUTCOMES:
correlation between diaphragm motion (mm) and forced vital capacity(ml) | 1 year
  using echography and FPT
correlation between diaphragm motion (mm) and inspiratory capacity (ml) | 1 year
  using echography and FPT
diaphragm thickness (mm) | 1 year
  using echography
correlation between diaphargm thickness and maximal inspiratory pressure (cmH20) | 1 year
  using echography and FPT

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Raymond Poincare, Garches, France

REFERENCES:
- [Derived] Fayssoil A, Nguyen LS, Stojkovic T, Prigent H, Carlier R, Amthor H, Bergounioux J, Zini J, Damez-Fontaine S, Wahbi K, Laforet P, Nicolas G, Behin A, Bassez G, Leturcq F, Ben Yaou R, Mansencal N, Annane D, Lofaso F, Orlikowski D. Determinants of diaphragm inspiratory motion, diaphragm thickening, and its performance for predicting respiratory restrictive pattern in Duchenne muscular dystrophy. Muscle Nerve. 2022 Jan;65(1):89-95. doi: 10.1002/mus.27432. Epub 2021 Oct 25. PMID 34618930